CLINICAL TRIAL: NCT02979743
Title: MRI-based Neuroimaging Predictors of Clinical Improvements Following Occupational Therapy (OT) or OT Puls Acupuncture and Massage Methods in Children With Cerebral Palsy
Brief Title: MRI-based Neuroimaging Predictors of Clinical Improvements Following Therapy in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Shenzhen Children's Hospital (Other Government); General Hospital of Ningxia Medical University (Other); Xijing Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Shaanxi Provincial People's Hospital (Other); Baoji Central Hospital (Other); Children's Hospital of Fudan University (Other); Hainan People's Hospital (Other); Zunyi Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016YFC0100300CP01
Record Dates: First submitted 2016-11-24; First posted 2016-12-02 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Brain Injury, Chronic; Cerebral Palsy
MeSH Terms: conditions — Brain Injury, Chronic; Cerebral Palsy | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Occupational therapy group (Placebo Comparator): The children worked with an occupational therapist for 4 hours a day for 5 days per week (totaling 40 hours) and initially concentrated on unilateral activities with the hemiplegic hand,and added bilateral activities during the second week.
  Interventions: Behavioral: Occupational therapy
- Occupational therapy puls acupuncture and massage methods (Active Comparator): The patients receive occupational therapy puls acupuncture and massage methods.
  Interventions: Behavioral: Occupational therapy; Other: Occupational therapy puls acupuncture and massage methods

INTERVENTIONS:
Behavioral: Occupational therapy
Other: Occupational therapy puls acupuncture and massage methods
  Arms: Occupational therapy puls acupuncture and massage methods

SUMMARY:
The aim of this study is to explore the relationship between brain MRI-metrics and hand function observed in children with cerebral palsy (CP),compared between baseline and the third month, and thus determine the early MRI-based neuroimaging predictor of clinical improvement following therapy in children with CP.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the commonest cause of neurological disability in children. The upper limbs are often affected, with significant hand involvement from an early age.There are various methods of treatment for CP children with hand function disability. However, there is a lack of effective methods to predict the prognosis.

This prospective cohort study will include children with occupational therapy (OT) or OT plus acupuncture and massage methods. Children with CP will be evaluated in terms of upper limb motor function using the manual ability classification system (MACS), fine motor function measure (FMFM). The Brain injuries of Children will be evaluated by MRI.

The aim of this study is to explore the relationship between brain MRI-metrics and hand function, compared between baseline and the third month, and thus determine the early MRI-based neuroimaging predictors of clinical improvements following therapy in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-18 years
* Spastic cerebral palsy
* The complete clinical and MRI data

Exclusion Criteria:

* previous acupuncture and massage methods
* botulinum toxin upper limb injections
* braces artifact, excessive motion, afraid to enter the MRI
* parents were not interested in the MRI sessions

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Fine motor function measure (scores) | Baseline
  It is acquired at baseline.
Fine motor function measure (scores) | The 3rd month
  It is acquired at 3 months later following therapy.

SECONDARY OUTCOMES:
Gross motor function measure and classification system (scores) | Baseline
  It is acquired at baseline.The system is a 5 level clinical classification system that describes the gross motor function of people with cerebral palsy on the basis of self-initiated movement abilities.
Gross motor function measure and classification system (scores) | The 3rd month
  It is acquired at 3 months later following therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu H, Jiang H, Wang X, Zheng J, Zhao H, Cheng Y, Tao X, Wang M, Liu C, Huang T, Wu L, Jin C, Li X, Wang H, Yang J. Treatment response prediction of rehabilitation program in children with cerebral palsy using radiomics strategy: protocol for a multicenter prospective cohort study in west China. Quant Imaging Med Surg. 2019 Aug;9(8):1402-1412. doi: 10.21037/qims.2019.04.04. PMID 31559169